CLINICAL TRIAL: NCT05702593
Title: The Immediate Effects of Hamstring Stretching Alone or Combined With Myofascial Release of the Hamstring Muscle on Masseter Muscle Activity, Pressure Pain Threshold, Active Mouth Opening, Hamstring Flexibility, and Forward Head Flexed Posture in Recreationally Active Participants: A Randomized, Double-Blind, Controlled Trial Study
Brief Title: Immediate Effects of Hamstring Stretching Alone or Combined With Myofascial Release
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, caglar soylu, Assistant Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36442
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hamstring Injury; Masseter; Myofascial Release; Stretching; Surface EMG; Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Muscle Stretching Exercises; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, double-blind, controlled trial. The participants were randomly (randomisation was performed using the website www.randomiser.org ) allocated to one of two groups
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Surface EMG Data Collection (Other): For each subject, EMG activity was recorded from the left and right superficial masseter muscles using a multichannel EMG device.The EMG recordings were obtained with three repetitions during mandibular rest, and maximal voluntary isometric contractions (MVIC) in intercuspation (isometry) pre and post-treatment. The EMG data were recorded for 5 seconds, and three trials with 30 seconds of rest between contractions were performed [Tosato, SENIAM].
  Interventions: Procedure: Static stretching; Procedure: Myofascial Release
- Pressure pain threshold (Other): The pressure pain threshold was measured using a mechanical pressure algometer (model Baseline® Dolorimeters - Fabrication Enterprises Inc) with a contact head of 1 cm2 area.
  Interventions: Procedure: Static stretching; Procedure: Myofascial Release
- Maximum Active Mouth Opening (MMO) (Other): A tape measure was used to determine the maximum active mouth opening (MMO).
  Interventions: Procedure: Static stretching; Procedure: Myofascial Release
- Hamstring Flexibility (Other): The Maximal Hip Flexion Active Knee Extension (MHFAKE) Test, which is an adapted active knee extension test, was performed to evaluate the hamstring flexibility of the participant.
  Interventions: Procedure: Static stretching; Procedure: Myofascial Release
- Tragus Wall Distance (Other): Tragus wall distance measurement was used to evaluate spinal mobility.
  Interventions: Procedure: Static stretching; Procedure: Myofascial Release
- Static stretching (Experimental): The participant was positioned supine for static stretching to be applied to the hamstring muscles
  Interventions: Procedure: Static stretching
- Myofascial Release (Experimental): For hamstring muscles, the participants were asked to assume a long sitting position on a firm, flat surface with their arms behind their backs and their body weight on their palms.
  Interventions: Procedure: Myofascial Release

INTERVENTIONS:
Procedure: Static stretching — The participant was positioned supine for static stretching to be applied to the hamstring muscles. The physiotherapist flexed the participant's hip to the point where resistance to the movement was first observed, with the knee extended.At this point, after waiting for 40 seconds, it was returned to the previous position. This application was made on both sides [Bretischwerdt]. The technique was repeated three times, with a 15-second rest interval between each repetition.
  Arms: Hamstring Flexibility; Maximum Active Mouth Opening (MMO); Pressure pain threshold; Static stretching; Surface EMG Data Collection; Tragus Wall Distance
Procedure: Myofascial Release — For hamstring muscles, the participants were asked to assume a long sitting position on a firm, flat surface with their arms behind their backs and their body weight on their palms. A foam roller was placed under the hamstring muscles and slowly moved the tuberositas ischii popliteus back and forth with pressure for 4 minutes.
  Arms: Hamstring Flexibility; Maximum Active Mouth Opening (MMO); Myofascial Release; Pressure pain threshold; Surface EMG Data Collection; Tragus Wall Distance

SUMMARY:
To assess the immediate effects of hamstring stretching alone or combined with myofascial release of the hamstring muscle on masseter muscle activity, pressure pain threshold, active mouth opening, hamstring flexibility, and forward head flexed posture in recreationally active participants. The young, healthy, recreationally active adults aged 18-25 years were included in the study. The participants were randomly separated into two groups of equal number. Static stretching alone was applied to one group and this was combined with myofascial release techniques (SSMR) for the other group. Masseter muscle activity was assessed using a NORAXON® surface electromyography device. Both pre-and post-intervention, mechanical pressure algometer was used to measure the pressure pain threshold, hamstring flexibility was evaluated using the maximum hip flexion and active knee extension test, the maximum mouth opening (MMO) was measured with the millimetric ruler, and forward flexed posture was evaluated using the tragus to wall distance test.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who had no previous hamstring injury
* Individuals had a Straight Leg Raise test <80°
* Individuals had a pressure-pain threshold difference between two symmetrical points not exceeding 2 kg/cm2
* Individuals who had no previous hamstring injury had no deviation during mouth opening and closing

Exclusion Criteria:

* acute low back pain or musculoskeletal pain in the lower extremities
* recent spinal surgery
* previous whiplash injury

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-01-22 (Actual); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
superficial masseter muscles EMG activity | 4 weeks
  For each subject, EMG activity was recorded from the left and right superficial masseter muscles using a multichannel EMG device.
Pressure pain threshold | 4 weeks
  The pressure pain threshold was measured using a mechanical pressure algometer (model Baseline® Dolorimeters - Fabrication Enterprises Inc) with a contact head of 1 cm2 area.The participant was positioned lying supine while the pressure pain threshold of the masseter muscle's central trigger point was assessed on both sides. Pressure was applied perpendicular to the masseter, gradually and continuously at a rate of about 1 kg/cm/s. The participants were requested to let the examiner know as soon as pain started to be felt. With a 2-min rest period between each experiment, three pressure pain threshold measures were taken. The average value of the three trials was calculated and used in the analysis.
Maximum Active Mouth Opening | 4 weeks
  A tape measure was used to determine the maximum active mouth opening (MMO). The participants were measured while laying flat on their back with the head resting on a table, the cervical spine in a neutral position, the knees slightly bent, and the upper limbs lying parallel to the torso. The subjects were instructed to open the mouth as wide as possible without inflicting discomfort. The distance between the upper and lower central incisors was measured and recorded in millimetres. For the primary analysis, the mean value of three trials was calculated.
Hamstring Flexibility | 4 weeks
  The Maximal Hip Flexion Active Knee Extension (MHFAKE) Test, which is an adapted active knee extension test, was performed to evaluate the hamstring flexibility of the participant. The subject was instructed to keep the hip in maximal flexion by clutching the thigh to the chest, with the hands holding the opposite elbows, and then to actively extend the knee until reaching the point of maximal tolerable stretch of the hamstring muscle or the point where pain was reported. The contralateral leg was fixed by the clinician. The angle of inclination of the mid-shin was measured at the endpoint of maximal stretch with the handheld inclinometer.
Tragus Wall Distance | 4 weeks
  Tragus wall distance measurement was used to evaluate spinal mobility. The participants were instructed to stand with their feet shoulder-width apart, and heels, hips, and shoulders against the wall. Then, before each measurement, the participants were asked to "stand with good posture, look straight ahead, and hold this position until the measurement is taken". The participants were then told to take a self-selected position for the head and neck that reflected their perception of "good posture". The distance between the tragus and the wall was measured and the participant was repositioned away from the wall before each measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Caglar Soylu, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided